CLINICAL TRIAL: NCT07234162
Title: A Phase 3, Open-Label, Randomized, Multinational Study to Investigate the Anti-tumor Efficacy of Golidocitinib Versus Investigator's Choice in Adult Patients With Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: A Phase 3 Multinational Study of Golidocitinib Versus Investigator's Choice in r/r PTCL (JACKPOT19)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022J0004
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; 10-propargyl-10-deazaaminopterin; Gemcitabine; belinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golidocitinib (Experimental)
  Interventions: Drug: Golidocitinib
- Investigator's Choice (Active Comparator)
  Interventions: Drug: Chidamide; Drug: Pralatrexate; Drug: Gemcitabine; Drug: Belinostat

INTERVENTIONS:
Drug: Golidocitinib — 150 mg, orally, once daily, with or without food, in a 21-day cycle
  Arms: Golidocitinib
Drug: Chidamide — 30 mg, orally, twice a week, with an interval of no less than 3 days in a 21-day cycle
  Arms: Investigator's Choice
Drug: Pralatrexate — 30 mg/m2, intravenous push, once weekly for 6 weeks in 7-week cycles
  Arms: Investigator's Choice
Drug: Gemcitabine — 1000 mg/m2, intravenous infusion, administered on Day 1, Day 8 and Day 15 of a 28-day cycle
  Arms: Investigator's Choice
Drug: Belinostat — 1000 mg/m2, intravenous infusion, administered once daily (QD) on Day 1 to Day 5 of a 21-day cycle
  Arms: Investigator's Choice

SUMMARY:
This is a phase 3, open-label, randomized, multinational study to evaluate the anti-tumor efficacy of golidocitinib versus investigator's choice in adult patients with relapsed/refractory peripheral T-cell lymphoma (r/r PTCL). This study will treat patients with pathologically confirmed PTCL who have relapsed after or been refractory/intolerant to at least one prior systemic treatment regimen(s).

ELIGIBILITY:
Inclusion Criteria:

* The participants should sign the ICF and be able to comply with the relevant requirement in the ICF and protocol
* Age ≥ 18 years
* ECOG 0-2 score, life expectancy ≥ 12 weeks
* Patients must have histologically confirmed peripheral T-cell lymphoma according to the World Health Organization classiﬁcation of lymphoma. Eligible subtypes are restricted to: PTCL-not otherwise specified, NOS (PTCL, NOS), Angioimmunoblastic T-cell lymphoma (AITL), anaplastic large-cell lymphoma ALK-positive (ALCL ALK+), anaplastic large-cell lymphoma ALK-negative (ALCL ALK-), Follicular T-cell lymphoma, or PTCL with T-follicular helper (TFH) phenotype (FTCL or PTCL-TFH), Enteropathy-associated T-cell lymphoma (EATL), Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), Natural killer/T-cell lymphoma (NK/TCL), Hepatosplenic T-cell lymphoma (HSTCL), Subcutaneous panniculitis-like T-cell lymphoma (SPTCL)
* Progressed on, were refractory to or intolerant to at least one line of prior standard systemic therapies assessed by investigator
* Adequate bone marrow reserve and organ system functions
* Willing to comply with contraceptive restrictions

Exclusion Criteria:

* Any of previous or current treatment prohibited by protocol
* Any unresolved > grade 2 drug-related adverse events
* Lymphoma involving central nervous system
* Any of serere cardiac or pulmonary abnormalities
* Disease condition requiring immunosuppressants, biologics, or NSAIDs
* Active infection
* Malignancy disease within five years
* Poorly controlled gastrointestinal disorder or inadequate absorption of medication
* Severe or poorly controlled systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the Independent Review Committee (IRC) according to Lugano 2014 | The time from the date of randomization to the date of first progressive disease, death due to any cause whichever occurred first. Approximately 4 years.

SECONDARY OUTCOMES:
Overall survival (OS) | The time from randomization to death due to any cause. Approximately 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao, Principal Investigator — Ruijin Hospital
Locations (50):
- China (36):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital & Institution, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Centeral Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Taiwan (8):
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center - Liouying Branch, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
- Thailand (6):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Mahidol University - Faculty of Medicine - Ramathibodi Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital - Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Prince of Songkla University-Faculty of Medicine, Hat Yai

IPD SHARING:
Plan to Share IPD: No